CLINICAL TRIAL: NCT02366975
Title: Effectiveness of Testosterone Replacement Therapy (TRT) on Prostatic Gland in Hypogonadal Patients Affected by Benign Prostatic Hyperplasia (BPH) and Metabolic Syndrome (MetS). Florence-PROTEST
Brief Title: TRT on BPH Hypoganadal MetS Patients. Florence-PROTEST
Acronym: PROTEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, Full Professor of Endocrinology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-003494-26
Record Dates: First submitted 2014-12-11; First posted 2015-02-19 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Hypogonadism
Keywords: BPH/LUTS; TRT; Metabolic Syndrome
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Hypogonadism; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eugonadal patients (No Intervention): Patients without hypogonadism has been enrollend but not randomized
- Hypogonadal patients A (Active Comparator): Patients with hypogonadism has been randomized to testosterone gel solution 2%
  Interventions: Drug: Testosterone gel 2%
- Hypogonadal patients B (Placebo Comparator): Patients with hypogonadism has been randomized to placebo solution gel
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Testosterone gel 2% — testosterone gel 2% (50mg/die).
  Other Names: tostran
  Arms: Hypogonadal patients A
Other: Placebo — placebo gel
  Arms: Hypogonadal patients B

SUMMARY:
There are many evidences in the literature showing that the metabolic syndrome (MetS) is associated with BPH / LUTS. There are also numerous evidence that hypogonadism is associated with both conditions, thus being one of the most probable pathogenetic factor underlying the association between MetS & BPH / LUTS.

Preliminary evidences from observational clinical studies have shown that treatment with testosterone replacement in hypogonadal patients with MetS reduces the symptoms of lower urinary tract symptoms (LUTS) associated with BPH. Preclinical studies performed by the investigators research group show in an experimental model of metabolic syndrome the occurrence of marked inflammation and tissue remodeling of the prostate gland, which is prevented by treatment with testosterone replacement (Vignozzi et al., 2012). There is therefore a need for a clinical trial to demonstrate the effect of treatment with testosterone replacement in reducing the inflammation of the prostate and its effectiveness in improving the symptoms related to inflammation in patients with prostatic BPH associated with metabolic syndrome and testosterone deficiency .

The aims of the present study is to evaluate the effectiveness of testosterone replacement therapy compared to placebo in reducing signs and symptoms of inflammation of the prostate and LUTS symptoms in hypogonadal patients with metabolic syndrome and BPH who are candidates for radical prostatectomy simple.

For this purpose both clinical (assessment of specific symptoms of prostatitis assessed by questionnaire National Institutes of Health Chronic Prostatitis Symptom Index, NIH-CPSI and assessment of the symptoms of LUTS and questionnaires International Prostate Symptom Score, IPSS), ultrasound (transrectal ultrasound evaluation of markers of prostatic inflammation: macrocalcifications, inhomogeneity etc.), biochemical (evaluation of inflammatory cytokines in the semen), urodynamic and histology (histomorphometric and immunohistochemical analysis of samples prostate derived from patients enrolled in the study or not treated with testosterone) scores will be performed. Along with the symptoms and clinical signs of prostate inflammation and LUTS, the effect of testosterone therapy or placebo on penile erection will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥ 18 years on the waiting list for simple prostatectomy for BPH
* Diagnosis of metabolic syndrome (AHA / NHLBI) defined by the presence of three or more of the following parameters: visceral obesity (waist circumference> or = 102 cm), fasting glucose (> or = 100 mg / dL) or a history of diabetes mellitus or treatment with antidiabetic drugs, high triglycerides (> or = 150 mg / dL) or treatment, high levels of blood pressure (BP> or = 130/85 mm Hg) or drug treatment and reduced levels of HDL cholesterol (<or = 40 mg / dL) or treatment.
* Diagnosis of prostatic inflammation defined by a score greater than 15 at the NIH-CPSI questionnaire
* Capacity to give consent for study participation, after being adequately informed of the aims, benefits, risks, time and motion of the study

Exclusion Criteria:

* Participation in another clinical trial;
* Previous diagnosis, presence or suspected malignancy of the prostate or breast cancer;
* PSA values10ng/mL
* Values of hematocrit ≥ 52%
* Use of 5alpha-reductase inhibitor drugs in the previous three months;
* Presence of a serious organic disease or mental diagnosed by a specialist psychiatrist (eg major depression medication) suspected on the basis of medical history and / or physical examination of the patient
* Presence of conditions that may affect the compliance to the study;
* Presence of severe allergy or hypersensitivity to study drug (active ingredient or excipients of the formulation);

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-11; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
NIH-CPSI | 6 months before surgery
  Evaluation in hypogonadal patients with both BPH and metabolic syndrome of the effectiveness of 6 months of treatment with testosterone compared with placebo in improving symptoms of prostatitis and the symptoms of LUTS
IPSS | 6 months before surgery
  Evaluation in hypogonadal patients with both BPH and metabolic syndrome of the effectiveness of 6 months of treatment with testosterone compared with placebo in improving symptoms of prostatitis and the symptoms of LUTS

SECONDARY OUTCOMES:
ultrasound prostate characteristics | 6 months before surgery
  Evaluation in hypogonadal patients with both BPH and metabolic syndrome of the effectiveness of 6 months of treatment with testosterone compared with placebo in improving
Immunohistological analysis of prostatic inflammation and gene expression of inflammatory markers on the prostate | 6 months before surgery
  Evaluation in hypogonadal patients with both BPH and metabolic syndrome of the effectiveness of 6 months of treatment with testosterone compared with placebo in improving
metabolic parameters | 6 months before surgery
  Evaluation in hypogonadal patients with both BPH and metabolic syndrome of the effectiveness of 6 months of treatment with testosterone compared with placebo in improving

CONTACTS AND LOCATIONS:
Overall Officials: mario maggi, Principal Investigator — University of Florence
Locations (2):
- Italy (2):
  - Ambulatori Medicina della Sessualità e Andrologia, Florence
  - Clinica Urologica - Azienda Ospedaliero-Universitaria Careggi, Florence

REFERENCES:
- [Result] Vignozzi L, Morelli A, Sarchielli E, Comeglio P, Filippi S, Cellai I, Maneschi E, Serni S, Gacci M, Carini M, Piccinni MP, Saad F, Adorini L, Vannelli GB, Maggi M. Testosterone protects from metabolic syndrome-associated prostate inflammation: an experimental study in rabbit. J Endocrinol. 2012 Jan;212(1):71-84. doi: 10.1530/JOE-11-0289. Epub 2011 Oct 18. PMID 22010203
- [Result] Cohen PG. Benign prostatic hyperplasia: the hypogonadal-obesity-prostate connection. Med Hypotheses. 2009 Aug;73(2):142-3. doi: 10.1016/j.mehy.2009.03.013. Epub 2009 Apr 24. PMID 19394149
- [Result] Filippi S, Vignozzi L, Morelli A, Chavalmane AK, Sarchielli E, Fibbi B, Saad F, Sandner P, Ruggiano P, Vannelli GB, Mannucci E, Maggi M. Testosterone partially ameliorates metabolic profile and erectile responsiveness to PDE5 inhibitors in an animal model of male metabolic syndrome. J Sex Med. 2009 Dec;6(12):3274-88. doi: 10.1111/j.1743-6109.2009.01467.x. Epub 2009 Sep 1. PMID 19732305
- [Result] Lotti F, Corona G, Colpi GM, Filimberti E, Degli Innocenti S, Mancini M, Baldi E, Noci I, Forti G, Adorini L, Maggi M. Elevated body mass index correlates with higher seminal plasma interleukin 8 levels and ultrasonographic abnormalities of the prostate in men attending an andrology clinic for infertility. J Endocrinol Invest. 2011 Nov;34(10):e336-42. doi: 10.3275/7855. Epub 2011 Jul 7. PMID 21738005